CLINICAL TRIAL: NCT04480333
Title: A Randomized, Placebo-controlled Study of the Safety, Tolerability and Pharmacokinetics of Inhaled Nanoparticle Formulation of Remdesivir (GS-5734) and in Combination With NA-831 in Healthy Volunteers
Brief Title: Safety, Tolerability and Pharmacokinetics of Inhaled Nanoparticle Formulation of Remdesivir (GS-5734) and NA-831
Acronym: NEUROSIVIR
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biomed Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NEUROSIVIR
Record Dates: First submitted 2020-07-13; First posted 2020-07-21 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Covid19; Corona Virus Infection; Severe Acute Respiratory Syndrome; Severe Acute Respiratory Infection; Severe Acute Respiratory Syndrome (SARS) Pneumonia; Severe Acute Respiratory Syndrome of Upper Respiratory Tract; Neurodegeneration; Neuroinflammatory Response
Keywords: Covid-19; Corona Virus Infection; Severe Acute Respiratory Syndrome; Severe Acute Respiratory Infection; Severe Acute Respiratory Syndrome (SARS) Pneumonia; Severe Acute Respiratory Syndrome of Upper Respiratory Tract; Neurodegeneration; Neuroinflammation; Cognitive decline
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Severe Acute Respiratory Syndrome; Pneumonia; Nerve Degeneration; Neuroinflammatory Diseases; Cognitive Dysfunction | interventions — remdesivir

STUDY DESIGN:
Intervention Model Description: The dose escalation given to healthy volunteers across the following cohorts:
  NA-831 cohorts:
  0.1 mg/kg NA-831, number of subjects N=2 and 2 subjects on placebos 0.2 mg/kg NA-831, number of subjects N=4 and 2 subjects on placebos 0.5 mg/kg NA-831, number of subjects N=4 and 2 subjects on placebos
  GS-5734 cohorts:
  1. mg/kg GS-5734, number of subjects N=2 and 2 subjects on placebos
  2. mg/kg GS-5734, number of subjects N=4 and 2 subjects on placebos
  4 mg/kg GS-5734, number of subjects N=4 and 2 subjects on placebos
  NA-831 plus GS-5734 cohorts:
  0.1 mg/kg NA-831 plus 1 mg/kg GS-5734, number of subjects N=2 and 2 subjects on placebos 0.2 mg/kg NA-831 plus 2 mg/kg GS-5734, number of subjects N=4 and 2 subjects on placebos 0.5 mg/kg NA-831 plus 4 mg/kg GS-5734, number of subjects N=4 and 2 subjects on placebos.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (12):
- Drug: NA-831 - 0.10 mg/kg (Experimental): 3 Subjects will take inhaled formulation of NA-831 once a day for 5 days
  Interventions: Drug: Drug: NA-831 - 0.10 mg/kg
- Comparable Placebo- 0.10 mg/kg (Placebo Comparator): 3 subjects will take inhaled formulation of placebo once a day for 5 days
  Interventions: Drug: Placebo- 0.10 mg/kg
- Drug: NA-831 - 0.20 mg/kg (Experimental): 6 Subjects will take inhaled formulation of NA-831 once a day for 5 days
  Interventions: Drug: Drug: NA-831 - 0.20 mg/kg
- Comparable Placebo- 0.20 mg/kg (Placebo Comparator): 3 subjects will take inhaled formulation of placebo once a day for 5 days
  Interventions: Drug: Placebo- 0.20 mg/kg
- Drug: GS-5734 - 1.00 mg/kg (Experimental): 3 Subjects will take inhaled formulation of GS-5734 once a day for 5 days
  Interventions: Drug: Drug: GS-5734 - 1.00 mg/kg
- Comparable Placebo- 1.00 mg.kg (Placebo Comparator): 3 Subjects will take inhaled formulation of GS-5734 once a day for 5 days
  Interventions: Drug: Placebo- 1.00 mg/kg
- Drug: GS-5734 - 2.00 mg/kg (Experimental): 6 Subjects will take inhaled formulation of GS-5734 once a day for 5 days
  Interventions: Drug: Drug: GS-5734 - 2.00 mg/kg
- Comparable Placebo - 2.00 mg/kg (Placebo Comparator): 3 Subjects will take inhaled formulation of GS-5734 once a day for 5 days
  Interventions: Drug: Placebo- 2.00 mg/kg
- Drugs: NA-831 (0.10 mg/kg) plus GS-5734 (1.00 mg/kg) (Experimental): 3 Subjects- will take inhaled formulation NA-831 (0.10 mg/kg) plus GS-5734 (1.00 mg/kg) once/day for 5 days
  Interventions: Combination Product: Drugs: NA-831 (0.10 mg/kg) plus GS-5734 (1.00 mg/kg)
- Placebo- 0.10- mg/kg placebo+1.00 mg mg/kg (Placebo Comparator): 3 Subjects - inhaled formulation of placebo once/day for 5 days
  Interventions: Combination Product: Placebo 0.10 mg + 1.00 mg/kg
- Drugs: NA-831( 0.20 mg/kg) + GS-5734 (2.00 mg/kg) (Experimental): 6 Subjects- inhaled formulation of NA-831 (0.20 mg/kg) + GS-5734 (2.00 mg/kg) once/day for 5 days
  Interventions: Combination Product: Drugs: NA-831 (0.20 mg/kg) plus GS-5734 (2.00 mg/kg)
- Placebo- 0.20 mg/kg + 2.00mg/kg (Placebo Comparator): 3 Subjects- inhaled formulation of placebo once/day for 5 days
  Interventions: Combination Product: Placebo 0.20 mg + 2.00 mg/kg

INTERVENTIONS:
Drug: Drug: NA-831 - 0.10 mg/kg — NA-831 in nanoparticle inhalation formulation
  Other Names: NA-831 is a neuroprotective and neurogenesis drug
  Arms: Drug: NA-831 - 0.10 mg/kg
Drug: Placebo- 0.10 mg/kg — Placebo in nanoparticle inhalation formulation
  Other Names: Placebo Comparator
  Arms: Comparable Placebo- 0.10 mg/kg
Drug: Drug: NA-831 - 0.20 mg/kg — NA-831 in nanoparticle inhalation formulation
  Other Names: NA-81 is a neuroprotective drug
  Arms: Drug: NA-831 - 0.20 mg/kg
Drug: Placebo- 0.20 mg/kg — Placebo in nanoparticle inhalation formulation
  Other Names: Placebo Comparator
  Arms: Comparable Placebo- 0.20 mg/kg
Drug: Drug: GS-5734 - 1.00 mg/kg — GS-5734 in nanoparticle inhaled formulation
  Other Names: GS-5734 (Remdesivir) is an antiviral drug
  Arms: Drug: GS-5734 - 1.00 mg/kg
Drug: Placebo- 1.00 mg/kg — Placebo in nanoparticle inhalation formulation
  Other Names: Placebo Comparator
  Arms: Comparable Placebo- 1.00 mg.kg
Drug: Drug: GS-5734 - 2.00 mg/kg — GS-5734 in nanoparticle inhaled formulation
  Other Names: GS-5734 (Remdesivir) is an anti-viral drug
  Arms: Drug: GS-5734 - 2.00 mg/kg
Drug: Placebo- 2.00 mg/kg — Placebo in nanoparticle inhaled formulation
  Other Names: Placebo Comparator
  Arms: Comparable Placebo - 2.00 mg/kg
Combination Product: Drugs: NA-831 (0.10 mg/kg) plus GS-5734 (1.00 mg/kg) — The combined NA-831 and GS-5734 are in nanoparticle inhaled formulation
  Other Names: Combination therapy of NA-831 a neuroprotective drug and GS-5734 an antiviral drug
  Arms: Drugs: NA-831 (0.10 mg/kg) plus GS-5734 (1.00 mg/kg)
Combination Product: Placebo 0.10 mg + 1.00 mg/kg — The combined placebo are in nanoparticle inhaled formulation
  Other Names: Placebo Comparator
  Arms: Placebo- 0.10- mg/kg placebo+1.00 mg mg/kg
Combination Product: Drugs: NA-831 (0.20 mg/kg) plus GS-5734 (2.00 mg/kg) — The combined NA-831 and GS-5734 are in nanoparticle inhaled formulation
  Other Names: Combination therapy of NA-831, a neuroprotective drug and GS-5734, an antiviral drug
  Arms: Drugs: NA-831( 0.20 mg/kg) + GS-5734 (2.00 mg/kg)
Combination Product: Placebo 0.20 mg + 2.00 mg/kg — Placebo 0.10 mg + 1.00 mg/kg
  Other Names: Placebo Comparator
  Arms: Placebo- 0.20 mg/kg + 2.00mg/kg

SUMMARY:
The clinical study is designed to evaluate the safety, tolerability and pharmacokinetics of inhaled nanoparticle nanoparticle formulation of Remdesivir (GS-5734) alone and in combination with NA-831 in 48 healthy volunteers.

DETAILED DESCRIPTION:
It has been discovered that SARS-CoV-2 viruses (Covid-19) can directly invade the nervous system of patients, instead of injuring the nervous system through the immune response. Neurotropism is one common feature of Covid-19. Such neuro-invasive propensity of Covid-19 has been documented almost for all the Beta-coronaviruses including SARS-CoV and MERS-CoV.

Increasing evidence suggests that infection with Sars-CoV-2 causes neurological deficits in a substantial proportion of affected patients. It was observed that patients surviving COVID-19 are at high risk for subsequent development of neurological disease and in particular Alzheimer's disease.

NA-831 is a new neuroprotective and neurogenesis drug that has been demonstrated its promising safety and efficacy in Phase 2A for the treatment of early onset of Alzheimer's disease. NA-831 in oral formulation is well tolerated NA-831 with no adverse effects. NA-831 in oral formulation exhibits predictable pharmacokinetics including dose-dependent exposure linearity and low variability.

Based on animal studies, NA-831 can provide effective interventions during the severe acute respiratory syndrome, and provide appropriate rehabilitation measures afterwards.

Remdesivir (GS-5734) intravenous formulation has been approved by the FDA under the emergency use authorization for potential treatment of severe cases of Covid-19.

It was found the upper respiratory tract is the most prevalent site of SARS-CoV-2 infection early in disease. Delivering drugs directly to the primary site of infection with a nebulizer, inhaled nanoparticle formulation may enable more targeted and accessible administration in non-hospitalized patients and potentially lower systemic exposure to the drug.

The study is designed to evaluate the safety, tolerability and pharmacokinetics of a new nanoparticle formulation of Remdesivir (GS-5734) and combination therapy with NA-831 in healthy volunteers.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Healthy adult volunteers, aged 21 to 50 years old, men or women.
2. Subjects negative for human immunodeficiency virus (HIV antibody screen), Hepatitis B virus surface Antigen (HBsAg) and Hepatitis C virus (HCV antibody screen).
3. Subjects who are willing to comply with the requirements of the study protocol, attend scheduled visits and make themselves available for the duration of the study with access to a consistent means of telephone contact.
4. Subjects who give written informed consent approved by the Internal Review Board governing the site.
5. Satisfactory baseline medical assessment as assessed by physical examination and a stable health status. Normal laboratory values must be within normal range of the assessing site or show minor variations that are deemed not clinically significant as judged by the Investigator and acceptable for study entry.
6. Accessible vein in the forearm for blood collection.
7. Female subjects of childbearing potential may be enrolled in the study if they have negative urine pregnancy tests on the day of screening and day of admission.
8. Female subjects of non-childbearing potential due to surgical sterilization (hysterectomy or bilateral oophorectomy or tubal ligation) or menopause.
9. Both male (if he has a partner of childbearing potential) and female subjects (of childbearing potential) must agree to use adequate and reliable contraceptive measures (e.g. spermicides, condoms, contraceptive pills, etc.) or practice abstinence throughout the duration of the study (up to 30 days post-dosing).

EXCLUSION CRITERIA:

1. Subject previously diagnosed with COVID-19 or had been issued with a quarantine order by the Center of Disease Control (CDC).
2. Presence of acute infection in the preceding 14 days, or presence of a temperature ≥ 100.0 ˚F (oral or tympanic temperature assessment), or acute symptoms of any severity on the scheduled date of admission.
3. History of severe drug and / or food allergies and / or known allergies to the trial product or its components.
4. Female subject who is pregnant or breast-feeding.
5. History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, , or immunosuppressive disorders.
6. Any neurological disease or history of significant neurological disorder (e.g. meningitis, seizures, multiple sclerosis, vasculitis, migraines, Guillain-Barré syndrome [genetic/congenital or acquired]).
7. Evidence of clinically significant anemia (HB < 10 g/dL) or any other significant active hematological disease, or having donated > 450 mL of blood within the past three (3) months.
8. Participation or planned participation in a study involving the administration of an investigational compound within the past four (4) months or during this study period.
9. Receipt of immunoglobulins and/or any blood products within nine (9) months of study enrolment or planned administration of any of these products during the study period.
10. Evidence of Hepatitis B or C or HIV by laboratory testing.
11. A positive test result for drugs of abuse (except a positive test result associated with prescription medication that has been reviewed and approved by the investigator) or alcohol at screening.
12. Administration of any licensed vaccine within 30 days before the first study vaccine dose.
13. Both male (if he has a partner of childbearing potential) and female subjects (of childbearing potential) who are unwilling to use adequate contraception or practice abstinence throughout the duration of the study (up to 84 days post-dosing).
14. Any condition that, in the opinion of the Investigator, would complicate or compromise the study or well-being of the subject.

    -

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-09-15 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants Experiencing any Treatment-Emergent Adverse Events | First dose date up to Day 30 Follow-up Assessment
  AEs will be assessed using Common Terminology Criteria for Adverse Events (CTCAE) V5.0
Proportion of Participants Experiencing any Treatment-Emergent Graded Laboratory Abnormalities | First dose date up to Day 30 Follow-up Assessment
  This will be assessed at various time points by clinical laboratory tests and vital signs.

SECONDARY OUTCOMES:
Maximum Concentration (Cmax) - Pharmacokinetic Assessment | 7 days
  Monitoring of the levels of drugs in subject sera at various time points to elucidate the maximum concentration (Cmax) of NA-831 and GS-5734 in human serum.
Time to Maximum Concentration (Tmax) - Pharmacokinetic Assessment | 7 days
  Monitoring of the levels of drugs in subject sera at various time points to elucidate the time to maximum concentration (Tmax) of NA-831 and GS-5734 in human serum
AUC calculated from time of administration to the last measurable concentration (AUC0-last) - Pharmacokinetic Assessment | 7 days
  Monitoring of the levels of drugs in subject sera at various time points to elucidate the area under the curve from time of administration to the last measurable of NA-831 and GS-5734
Area Under the Curve Extrapolated to Infinity (AUC0-∞) | 7 days
  Monitoring of the levels of drugs in subject sera at various time points to elucidate the area under the curve extrapolated to infinity (AUC0-∞) of NA-831 and GS-5734
Half-Life (t1/2) - Pharmacokinetic Assessment | 7 days
  Monitoring of the levels of drugs in subject sera at various time points to elucidate the half-life (t1/2) of NA-831 and GS-5734 in human serum.
Volume of Distribution (Vd) - Pharmacokinetic Assessment | 7 days
  Monitoring of the levels of drugs in subject sera through various time points to elucidate the volume of distribution (Vd) of NA-831 and GS-5734 in human serum.
Clearance [CL] - Pharmacokinetic Assessment | 7 days
  Monitoring of the levels of drugs in subject sera through at various time points to elucidate clearance [CL] of NA-831 and GS-5734 in human serum.

CONTACTS AND LOCATIONS:
Overall Officials: Lloyd Tran, PhD, Study Director — Biomed Industries, Inc.
Locations (1):
- Coronavirus Research Institute, Sunnyvale, California, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to share the Study Protocol
Supporting Information: Study Protocol
Time Frame: 90 days after the completion of the study
Access Criteria: to be determined